CLINICAL TRIAL: NCT06257498
Title: Upright Open MRI for Brain Imaging in Children - a Pilot Study
Acronym: Heads-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20DI001
Record Dates: First submitted 2024-01-23; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Brain Tumor
Keywords: Upright open scanner; MRI; Magnetic Resonance Imaging
MeSH Terms: conditions — Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI upright open scanner (Other): All participants will undergo MRI scanning in the dedicated open upright 0.5T MRI research MRI scanner , with parents or guardian in attendance if desired, and with their own choice of music or video during the scan.
  Immediately following the MRI scan we will collect information relating to their experience of the upright scanner using an age-appropriate questionnaire, based on similar questionnaires that we have used for paediatric MRI studies previously. A photograph of the upright MRI room will be used to prompt this discussion. The parent or carer may also be involved in prompting the child's responses.
  We will also collect the views of the parent / carer using a questionnaire.
  Interventions: Procedure: MRI scan

INTERVENTIONS:
Procedure: MRI scan — MRI scan on open scanner and some questionnaires

SUMMARY:
PRIMARY OBJECTIVE To establish feasibility and acceptability of diagnostic brain MRI in young children for specified indications using an upright MRI system without sedation or anaesthesia.

SECONDARY OBJECTIVES To establish how young children who undergo brain MRI using upright MRI view the experience To establish how parents / carers of young children who undergo brain MRI using the upright MRI view the experience for their child and for themselves.

To establish how image quality compares between brain MRI using the upright MRI scanner and the standard MRI scanner used in clinical practice.

DETAILED DESCRIPTION:
Study Design Feasibility study collecting data on image quality and experience of upright open MRI scanning (performed in addition to standard clinical MRI scan), and comparing outcome measures to standard supine MRI scans, in children referred for clinical MRI scanning for (i) symptoms or signs suggestive of brain tumour and (ii) symptoms or signs suggestive of shunt blockage in children with a ventriculoperitoneal (VP) shunt Study Participants Participants that have been referred for brain MRI for symptoms and signs suggestive of brain tumour or who have known VP shunts with a clinical suspicion of shunt dysfunction. 20 participants in total, aiming for an even split between these two groups but will be flexible based on the local clinical case load.

Planned Size of Sample (if applicable) 20 young school-aged children (5 to 10 years) referred for brain MRI at NUH. The child participant's parents will be simultaneously recruited

ELIGIBILITY:
Inclusion Criteria:

* Referred for clinical brain MRI scan for either:

Symptoms and signs suggestive of brain tumour, or Known VP shunts with a clinical suspicion of shunt dysfunction Parental consent and child's agreement to participate

Inclusion criteria for the adult participants:

Parent / carer of a child participant

Exclusion Criteria:

* Contra-indication to MRI scans Programmable VP shunt requiring re-programming after the research MRI Unable to sit upright unsupported Focal intracranial signs such that a targeted MRI protocol would be required (e.g. focal seizures, focal neurology, visual impairment, pituitary dysfunction).

Exclusion criteria for the adult participants:

Contra-indication to being in the scan room

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
MRI scan feasibility and image quality rating (by neuroradiologists) . | within 4 weeks of diagnostic MRI scan
  To establish feasibility and acceptability of diagnostic brain MRI in young children for specified indications using an upright MRI system without sedation or anaesthesia. Two experienced neuroradiologists blinded to patient and scanner will assess image quantity and motion artifact on each scan and rating image quality on a five point likert scale.Exams classified as 3, 4, or 5 "good", "very good" and " excellent" are considered diagnostic. The primary acceptability endpoint is defined as: 'more than 75% of child participants reporting a positive experience of the upright open MRI scan'.

SECONDARY OUTCOMES:
Scan acceptability- child questionnaires before and after each scan | all the questionnaires will be completed on the study day visit for the research scan, this will be within four weeks of the diagnostic clinical scan
  To establish how young children who undergo brain MRI using upright MRI view the experience using age appropriate questionaires.The primary acceptability endpoint is defined as: 'more than 75% of child participants reporting a positive experience of the upright open MRI scan'.
Scan acceptability - patient /Carer questionaire before and after each scan. | all the questionnaires will be completed on the study day visit for the research scan, this will be within four weeks of the diagnostic clinical scan
  To establish how parents / carers of young children who undergo brain MRI using the upright MRI view the experience for their child and for themselves using questionaires. The primary acceptability endpoint is defined as: 'more than 75% of participants reporting a positive experience for their child of the upright open MRI scan'.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Dineen, prof, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marshall SP, Smith MS, Weinberger E. Perceived anxiety of pediatric patients to magnetic resonance. Clin Pediatr (Phila). 1995 Jan;34(1):59-60. doi: 10.1177/000992289503400114. No abstract available. PMID 7720333
- [Background] Chou IJ, Tench CR, Gowland P, Jaspan T, Dineen RA, Evangelou N, Abdel-Fahim R, Whitehouse WP, Constantinescu CS. Subjective discomfort in children receiving 3 T MRI and experienced adults' perspective on children's tolerability of 7 T: a cross-sectional questionnaire survey. BMJ Open. 2014 Oct 15;4(10):e006094. doi: 10.1136/bmjopen-2014-006094. PMID 25320001
- [Background] Hallowell LM, Stewart SE, de Amorim E Silva CT, Ditchfield MR. Reviewing the process of preparing children for MRI. Pediatr Radiol. 2008 Mar;38(3):271-9. doi: 10.1007/s00247-007-0704-x. Epub 2007 Dec 15. PMID 18084752
- [Background] Carter AJ, Greer ML, Gray SE, Ware RS. Mock MRI: reducing the need for anaesthesia in children. Pediatr Radiol. 2010 Aug;40(8):1368-74. doi: 10.1007/s00247-010-1554-5. Epub 2010 Feb 26. PMID 20186541
- [Background] de Amorim e Silva CJ, Mackenzie A, Hallowell LM, Stewart SE, Ditchfield MR. Practice MRI: reducing the need for sedation and general anaesthesia in children undergoing MRI. Australas Radiol. 2006 Aug;50(4):319-23. doi: 10.1111/j.1440-1673.2006.01590.x. PMID 16884416